CLINICAL TRIAL: NCT03269682
Title: Prevalence of Contrast Enhancement of the Oculomotor Nerve on 3D PD T1 MRI Sequence in Patients With Ophthalmoplegia
Acronym: 3D-III
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: FHN_2017_4
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Ophthalmoplegia
MeSH Terms: conditions — Ophthalmoplegia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 3D PD T1 MRI sequence — After MRI has been performed (about 5 minutes of additional time compared to the usual sequences), a double reading of the MRI will be performed by two radiologists (1 experienced and 1 junior).

SUMMARY:
Oculomotor nerve (third cranial nerve or "III") palsy is a relatively frequent cause of consultation in ophthalmology.

It may reveal a life-threatening pathology such as aneurysm rupture, pituitary apoplexy, and therefore need imaging in emergency. Apart from few extreme emergency situations, MRI of the oculomotor tract is the first-line examination required. In our usual clinical practice, we noticed in several patients unusual contrast enhancement within the oculomotor nerve on T1 sequence with gadolinium injection, observed in various locations along the nerve path (cavernous and/ or intra-orbital segment).

This contrast enhancement, could confirm the nerve impairment This study aims to analyse the efficiency of a new sequence 3D PD T1 which isotropic spatial resolution less than 1mm, not yet described in the literature, to depict this enhancement.

In patients with ophthalmoplegia involving probably the third cranial nerve, disclosing this MRI sign could help (i) to confirm the involvement of the oculomotor nerve and eliminate differential diagnoses such as myasthenia (ii) to orientate the etiological diagnosis (inflammatory or ischemic origin). This new sequence 3D PD T1 sequence focused on the III could thus be systematically included in the usual MRI protocol.

ELIGIBILITY:
Inclusion Criteria:

- Ophthalmoplegia whatever the clinical form (unilateral or not, isolated or not, sudden or progressive onset)

Exclusion Criteria:

-Absolute contraindication to MRI or injection of contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ophtalmoplegia
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Contrast enhancement of the oculomotor nerve on 3D PD T1 MRI sequence (presence or absence, determined by a radiologist) | Baseline
  A double separate reading of the imaging will be carried out by an experienced radiologist and a junior radiologist on anonymized MRIs, with no access to clinical elements and interpretation of the other radiologist. In case of discrepancy between the radiologists, the final decision will be made by a third experienced radiologist under the same conditions (no access to clinical data, no access to the other evaluations).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided